CLINICAL TRIAL: NCT03291106
Title: Cohort Study of Universal Screening for Lynch Syndrome in Chinese Patients of Endometrial Cancer
Brief Title: Study of Universal Screening for Lynch Syndrome in Chinese Patients of Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EC-LYNCH
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: immunohistochemical staining — immunohistochemical staining for MLH1, MSH2, MSH6 and PMS2
Diagnostic Test: tests of microsatellite instability — microsatellite instability in tissues of endometrial cancer
Diagnostic Test: clinical criteria of Lynch syndromes — Amsterdam I or II criteria and Bethesda criteria
Diagnostic Test: sequencing for mismatch repair genes — next-generation sequencing, Sanger method or qPCR for mismatch repair genes (MLH1, MSH2, MSH6, PMS2, and EPCAM)

SUMMARY:
In patients diagnosed as endometrial cancer by thorough pathologic examinations, Lynch syndromes are screened by (1)immunohistochemical staining (for MLH1, MSH2, MSH6 and PMS2), (2) tests of microsatellite instability and (3) clinical criteria (Amsterdam I or II criteria and Bethesda criteria). For patients with any suspicious discoveries of Lynch syndromes from aforementioned screening methods, a molecular diagnosis with next-generation sequencing for mismatch repair genes (MLH1, MSH2, MSH6, PMS2, and EPCAM) is given to confirm Lynch syndromes. For patients of Lynch syndromes and endometrial cancer, relatives of blood lineage are tested by Sanger method or qPCR to find out carriers of mutation genes of Lynch syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Survivals of endometrial cancer

Exclusion Criteria:

* Metatatic malignacies to uterine
* Leiomyosarcoma of uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens with definite diagnosis of endometrial cancer, including type I and type II endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of Lynch syndromes in endometrial cancer | 2 years
  Proportions of patients carrying mismatch repair gene in endometrial cancer

SECONDARY OUTCOMES:
Reliability of immunohistochemical staining for screening Lynch syndromes | 2 years
  Sensitiviy and specitiviy of immunohistochemical staining for screening Lynch syndromes
Reliability of microsatellite instability for screening Lynch syndromes | 2 years
  Sensitiviy and specitiviy of microsatellite instability for screening Lynch syndromes
Reliability of clinical criteria for screening Lynch syndromes | 2 years
  Sensitiviy and specitiviy of clinical criteria for screening Lynch syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Distributions of specific mutation genes of Lynch syndromes will be available for other researches by officially published papers.
Supporting Information: CSR

REFERENCES:
- [Derived] Chao X, Li L, Wu M, Ma S, Tan X, Zhong S, Bi Y, Lang J. Comparison of screening strategies for Lynch syndrome in patients with newly diagnosed endometrial cancer: a prospective cohort study in China. Cancer Commun (Lond). 2019 Jul 15;39(1):42. doi: 10.1186/s40880-019-0388-2. PMID 31307542